CLINICAL TRIAL: NCT04031196
Title: Ultrasound-guided Quadratus Lumborum Block Versus Transversus Abdominis Plane Block in Children Undergoing Laparoscopic Appendicectomy: A Randomized Clinical Study
Brief Title: Quadratus Lumborum Block Versus Transversus Abdominis Plane Block in Children Undergoing Laparoscopic Appendicectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Shereen Elsayed Abd Ellatif, lecturer of anesthesia and surgical intensive care, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 5504-16-9-2018
Record Dates: First submitted 2019-07-17; First posted 2019-07-24 (Actual); Last update posted 2020-08-07 (Actual); Status verified 2020-08

CONDITIONS: Children; Appendicitis
Keywords: Pediatric; Quadratus Lumborum; regional anesthesia
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Intervention Model Description: 34 patients randomly allocated into two equal groups 17 patients in each group: Quadratus Lumborum Block" QLB group": ultrasound-guided QLB type 2 with 0.5ml/kg of 0.25% levobupivacaine local anesthetic was done to patients.
  and Transversus Abdominis Plane Block group (TAP block): ultrasound-guided TAP block with 0.5ml/kg of 0.25% levobupivacaine local anesthetic was done to patients.
Who Masked: Participant, Care Provider
Masking Description: the participants were masked for the type of regional anesthesia given the care provider was blind to the type of the regional block given to the patient and he was asked to assess the visual analogue scale score, first time of rescue analgesia, the total dose of rescue analgesia given and postoperative side effects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QLB group, Quadratus Lumborum Block group (Active Comparator): the patient placed in the lateral decubitus position, the low-frequency convex probe of Sonosite M Turbo ultrasonography was placed in the anterior axillary line midway between subcostal margin and iliac crest to identify the abdominal muscle layers, then the probe was moved to the posterior axillary line to visualize the quadratus lumborum muscle attached to the transverse process of the L4, With the psoas major muscle placed anteriorly, the erector spinae muscle posteriorly, a 22-gauge, 80 mm needle was inserted in-plane into the posterior aspect of QL muscle (between quadratus lumborum and erector spinae muscle), and then 0.5ml/kg of 0.25% levobupivacaine local anesthetic was injected behind the muscle as a bolus dose. The block was performed bilaterally.
  Interventions: Procedure: QLB
- TAP block group,Transversus Abdominis Plane Block group (Active Comparator): patient placed in the supine position, a linear multifrequency 6-13 MHz probe of Sonosite M Turbo ultrasonography was placed posterior to the midaxillary line at the midpoint between the inferior costal margin and the iliac crest, a 22-gauge, 50 mm needle was placed using an in-plane technique between the internal oblique and transversus abdominis muscle then local anesthetic was injected in a bolus dose 0.5ml/kg of 0.25% levobupivacaine, the block was done bilaterally.. after ultrasound Identification of the plane between the internal oblique and transversus abdominis muscle,
  Interventions: Procedure: TAP block

INTERVENTIONS:
Procedure: QLB — QLB type 2 approach
  Arms: QLB group, Quadratus Lumborum Block group
Procedure: TAP block — classic TAP block approach
  Arms: TAP block group,Transversus Abdominis Plane Block group

SUMMARY:
QL block has been recently described for chronic pain following abdominal hernia repair, and for postoperative analgesia following abdominal surgery as it leads to complete pain relief in the dermatomal area from (T6 - L1). Theoretically, QL blocks might give better and longer-lasting analgesia compared to the US-guided anterior TAP block due to a spread to the thoracic paravertebral space and sympathetic nerves in the thoracolumbar fascia, so visceral afferent pathways to the medulla can be blocked.

DETAILED DESCRIPTION:
Recently, the laparoscopic technique has been successfully used for many pediatric surgical cases. The laparoscopic appendicectomy is favored over the traditional open method, as it has a lower incidence of postoperative surgical complications and faster recovery to normal daily activities. Although it is considered as minimally invasive surgery, patients may require hospitalization for over 24 hours following laparoscopic appendicectomy, and postoperative pain which is caused by the surgical wound and visceroperitonitic pain as a result of peritoneal inflammation and infection, may extend the length of hospital stay.

Regional anesthesia techniques are commonly enhanced for pain management in pediatric surgical procedure as they decrease parenteral opioid requirements and improve patient-parent satisfaction [6].

The Transversus Abdominis Plane (TAP) block was first described in 2004 by McDonnell et al. using anatomical landmark guidance, and ultrasound-guided technique was later popularized by Hebbard et al. TAP block is aiming to block sensory nerves that course between the transversus abdominis and internal oblique muscles and supply the anterior abdominal wall, where local anesthetic is injected into the transversus abdominis fascial plane. Many clinical studies have reported the efficacy of TAP block in providing adequate postoperative analgesia for lower abdominal surgery.

Quadratus Lumborum block was initially described by R.Blanco as an abstract at the annual European Society of Regional Anaesthesia (ESRA) congress in 2007, where the local anesthetic (LA) was injected in the anterolateral aspect of the QL muscle (type 1 QL block). Later, J. Børglum used posterior transmuscular approach by detecting Shamrock sign and injecting the LA in the anterior aspect of the QL (type 3 QL block). Recently, R. Blanco described another approach by injecting the LA in the posterior aspect of the QL muscle (type 2 QL block), which may be easier and safer as the LA is injected in a more superficial plane, so the risk of intra-abdominal complications and lumbar plexus injuries is reduced. And finally the intramuscular QL block (type 4 QL block), the local anesthetic is injected directly into the QL muscle.

We hypothesize that ultrasound-guided QL block will be more superior than or equal to TAP block in providing postoperative analgesia for children undergoing laparoscopic appendicectomy.

ELIGIBILITY:
Inclusion Criteria:

* parent and patient acceptance,
* Children 7-12 years old,
* 20-35kg bodyweight,
* ASA I-II,

  * and scheduled for Laparoscopic appendicectomy

Exclusion Criteria:

* Patients refusing regional anesthesia,
* those with bleeding disorders,
* skin lesion at the needle insertion site,
* sepsis,
* liver disease,
* peritonitis,
* and emergency cases

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
changes in intraoperative mean arterial blood pressure (MAP) values | at base line (To), 3 minutes(min) after induction of general anesthesia, 10 min after intubation (immediately before performing the block (T1)), 15 min after performing the block (T2),and intraoperative values every 15 min till the end of surgery(T3)
  (mm Hg)
changes in intraoperative heart rate (HR) values | at base line (To), 3 minutes(min) after induction of general anesthesia, 10 min after intubation (immediately before performing the block (T1)), 15 min after performing the block (T2),and intraoperative values every 15 min till the end of surgery(T3)
  (beats/minute)
changes in the degree of pain perception by patient | Patients were assessed in the immediate post operative period and then at 2 hour(h), 4h, 6h , 8h , 12 h, 18 h and at 24 hours postoperative for the quality of analgesia
  measured by visual analogue scale(VAS), The patient was trained to report the level of pain on VAS scale from 0 to 10 (where 0 indicates no pain and 10 indicates the most severe pain).

SECONDARY OUTCOMES:
total intraoperative fentanyl consumption | during the time of the surgical procedure
  measured by μg /kg
1st time of rescue analgesics | during the first postoperative 24 hours
  minute
total amount of rescue analgesic consumed | in the first postoperative 24 hours
  mg/kg
post operative nausea and vomiting | in the first postoperative 24 hours
  by number of patients complained of these side effects
degree of patient and parent satisfaction | at the end of the first postoperative 24 hours
  5-point scale assessment (satisfied or completely satisfied, not satisfied nor dissatisfied, dissatisfied, completely dissatisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Shereen E Abd Ellatif, MD, Principal Investigator — Anesthesia and Surgical Intensive Care Department, Faculty of medicine, Zagazig University; Fatma M Ahmed, MD, Study Director — Anesthesia and Surgical Intensive Care Department, Faculty of medicine, Zagazig University
Locations (1):
- Faculty of medicine, zagazig university, Zagazig, Elsharqya, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All the IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: the IPD and any additional supporting information will become available starting 6 months after publication
Access Criteria: by contacting the study director

REFERENCES:
- [Background] Gupta V, Yadav SK, Dean E, Vincent P, Walid F, Al Said A. Paediatric laparoscopic orchidopexy as a novel mentorship: Training model. Afr J Paediatr Surg. 2013 Apr-Jun;10(2):117-21. doi: 10.4103/0189-6725.115035. PMID 23860059
- [Background] Bharti N, Kumar P, Bala I, Gupta V. The efficacy of a novel approach to transversus abdominis plane block for postoperative analgesia after colorectal surgery. Anesth Analg. 2011 Jun;112(6):1504-8. doi: 10.1213/ANE.0b013e3182159bf8. Epub 2011 Apr 5. PMID 21467560
- [Background] Siddiqui MR, Sajid MS, Uncles DR, Cheek L, Baig MK. A meta-analysis on the clinical effectiveness of transversus abdominis plane block. J Clin Anesth. 2011 Feb;23(1):7-14. doi: 10.1016/j.jclinane.2010.05.008. PMID 21296242
- [Background] Kadam VR. Ultrasound-guided quadratus lumborum block as a postoperative analgesic technique for laparotomy. J Anaesthesiol Clin Pharmacol. 2013 Oct;29(4):550-2. doi: 10.4103/0970-9185.119148. PMID 24249997
- [Background] Tupper-Carey DA, Fathil SM, Tan YK, Kan YM, Cheong CY, Siddiqui FJ, Assam PN. A randomised controlled trial investigating the analgesic efficacy of transversus abdominis plane block for adult laparoscopic appendicectomy. Singapore Med J. 2017 Aug;58(8):481-487. doi: 10.11622/smedj.2016068. Epub 2016 Apr 8. PMID 27056207
- [Background] Murouchi T. Quadratus lumborum block intramuscular approach for pediatric surgery. Acta Anaesthesiol Taiwan. 2016 Dec;54(4):135-136. doi: 10.1016/j.aat.2016.10.003. Epub 2016 Dec 9. No abstract available. PMID 27939905
- [Background] Visoiu M, Yakovleva N. Continuous postoperative analgesia via quadratus lumborum block - an alternative to transversus abdominis plane block. Paediatr Anaesth. 2013 Oct;23(10):959-61. doi: 10.1111/pan.12240. Epub 2013 Aug 9. PMID 23927552
- [Background] Blanco R, Ansari T, Riad W, Shetty N. Quadratus Lumborum Block Versus Transversus Abdominis Plane Block for Postoperative Pain After Cesarean Delivery: A Randomized Controlled Trial. Reg Anesth Pain Med. 2016 Nov/Dec;41(6):757-762. doi: 10.1097/AAP.0000000000000495. PMID 27755488